CLINICAL TRIAL: NCT01487343
Title: A Pilot Study to Identify Patient Factors Impacting Adherence to Oral Chemotherapy
Brief Title: Patient Factors Impacting Adherence to Oral Chemotherapy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-194
Record Dates: First submitted 2011-11-30; First posted 2011-12-07 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer; Gastrointestinal Cancer
Keywords: Oral Chemotherapy; capecitabine; questionnaire; breast; gastric; 11-194
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- breast or gastrointestinal cancer pts taking capecitabine: This is a mixed-methodology pilot study of patients currently taking oral chemotherapy for breast or gastrointestinal cancer. The quantitative portion of the study consists of self-report questionnaires assessing adherence, beliefs about medications, side effect experience, self-efficacy, and satisfaction with patient education; the qualitative portion is an interview guided by two open-ended questions.
  Interventions: Behavioral: questionnaire and interview

INTERVENTIONS:
Behavioral: questionnaire and interview — Interviews will be conducted with the first 10 participants who agree to be interviewed (or until data saturation is reached). Self-report questionnaires assessing adherence, beliefs about medications, side effect experience, self-efficacy, and satisfaction with patient education; the qualitative portion is an interview guided by two open-ended questions. Data will be collected approximately 2 weeks - 6 months (2 - 24 weeks) after being prescribed capecitabine.

SUMMARY:
The purpose of this study is to identify what makes it easier and what makes it harder to take oral chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary breast cancer or gastrointestinal cancer
* Currently prescribed capecitabine
* Age 21 years or older
* Able to understand written and oral English

Exclusion Criteria:

* Major psychopathology or cognitive impairment likely in the judgment of the research staff to interfere with the participation or completion of the protocol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2011-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
adherence to oral chemotherapy | 1 year
  Participation in the study entails completion of five short questionnaires related to the medication adherence (Medication Adherence Questionnaire), beliefs about medication (Beliefs about Medications Questionnaire), side effect experience (Frequency, Intensity, and Burden of Side Effects Rating), self-efficacy (Self-efficacy for Appropriate Medication Use) and satisfaction with medication information (Satisfaction with Information about Medicines Scale) as well as a demographic and treatment data sheet.

SECONDARY OUTCOMES:
improve the care of patients | 1 year
  Participation in the study entails completion of five short questionnaires related to the medication adherence (Medication Adherence Questionnaire), beliefs about medication (Beliefs about Medications Questionnaire), side effect experience (Frequency, Intensity, and Burden of Side Effects Rating), self-efficacy (Self-efficacy for Appropriate Medication Use) and satisfaction with medication information (Satisfaction with Information about Medicines Scale) as well as a demographic and treatment data sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Ginex, EdD, RN, OCN, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/